CLINICAL TRIAL: NCT06683664
Title: Human Papillomavirus Vaccine Integrated Service Implementation Research in Cameroon
Brief Title: HPV Vaccine Integrated Service Implementation Research in Cameroon
Acronym: HPV-PASSREV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Services International (Other)
Collaborators: Fobang Institutes for Innovations in Science and Technology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1861.2.2024; GAVI100001663 (Other Grant/Funding Number: Gavi, The Vaccine Alliance)
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Papillomavirus Vaccines; HPV Vaccinations; HPV Vaccines; HPV Vaccine Acceptability; HPV Vaccine Attitudes; HPV Vaccine Knowledge; Adolescent Health; Adolescent Health Services
Keywords: Implementation Science; Cameroon; Implementation Research; Mixed Methods

STUDY DESIGN:
Intervention Model Description: Cluster-assigned intervention treatment with concurrent comparison clusters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated health service delivery for very young adolescents (Experimental): The intervention will be implemented in 90 non-randomly selected health facilities and their catchment areas located in the North and Far North Regions of Cameroon. In intervention areas, the intervention (a complex, supply- and demand-side implementation model with the primary objective of increasing access to HPV vaccination and other health services for very young adolescents girls and boys [aged 9-13 years]) will be developed in the study's phase 1, a rapid formative phase. It is anticipated that the intervention will include supply- and demand-side components, such as household mobilization by community health workers engaged through the exiting Programme d'Accès aux Services de Santé de la Reproduction (PASSR), strengthened linkages between households and health facilities, and routinized HPV and adolescent health service delivery within communities.
  Interventions: Other: Integrated health service delivery for very young adolescents
- Standard of care (No Intervention): 90 non-randomly selected health facilities and their catchment areas supported by the Programme d'Accès aux Services de Santé de la Reproduction (PASSR) have been selected as concurrent comparison areas. These sites will conduct HPV vaccination (and other other adolescent health service delivery) through the standard-of-care procedures.

INTERVENTIONS:
Other: Integrated health service delivery for very young adolescents — The proposed HPV-PASSREV intervention will aim to increase adolescent-centered access to HPV vaccination and other very young adolescent health services through an integrated, routine, community-based delivery model that incorporates household mobilization efforts with enhanced service delivery at the health facility and community levels.
  Arms: Integrated health service delivery for very young adolescents

SUMMARY:
The goal of this implementation research study is to understand whether a package of community-based interventions can increase access to and uptake of the human papillomavirus (HPV) vaccine among very young adolescent girls and boys in the North and Far North Regions of Cameroon. The main questions this study aims to answer are:

* Can a package of community-based interventions increase delivery of routine HPV vaccination to boys and girls aged 9-13 in Cameroon's North and Far North Regions?
* What is the acceptability, feasibility, cost, and potential for maintenance and scale of an integrated health intervention to deliver routine HPV vaccination in Cameroon?

To evaluate the effectiveness of the intervention, researchers will compare HPV vaccination within regions where the new intervention model is being implemented (intervention areas) to regions where the new routine HPV vaccination delivery model is not being implemented (comparison areas) for approximately 1 year before the new intervention model is implemented and for approximately 9 months after the start of implementation to compare changes over time and between intervention and comparison areas.

The study will evaluate the effect of the intervention on HPV vaccination delivery using routine health facility data.

To understand acceptability, feasibility, implementation, and potential for scale, the study will enroll participants including health officials and providers, adolescents girls receiving HPV vaccination and other services in intervention areas, and their parents/caregivers. The study will be conducted in two phases, with the first phase focused on gathering formative data through interviews with key informants. This data will be used to inform the design of the intervention, which will be implemented and evaluated in phase 2. Only phase 1 of this study protocol has been currently approved.

In phase 1, key informant interview participants will be asked to participate in a an interview to discuss HPV vaccination services and their perspectives on how to integrate HPV vaccination within existing community-based and health facility structures and programs. Key informants will include government officials, health program implementers, representatives from non-government organizations working on HPV vaccine delivery, and healthcare providers, as well as community leaders including school and religious leaders.

DETAILED DESCRIPTION:
Introduction Cervical cancer is a leading cause of cancer among women in Cameroon. Vaccinating very young adolescent girls and boys is the most effective long-term strategy to reduce its risk. Despite the introduction of the human papillomavirus (HPV) vaccine in Cameroon in 2020, the vaccination program has faced substantial challenges, including widespread vaccine hesitancy and low awareness of the vaccine. As a result, an initial approach focusing on school-based vaccination was shifted to routine, health facility-based distribution. Integrating HPV vaccinations into existing health platforms that reach very young adolescents and their caregivers presents an opportunity to improve the effectiveness, acceptability, and feasibility of routine, community-based HPV vaccination in Cameroon. Implementation research is needed to evaluate the effectiveness of such integrated service delivery approaches, contributing to more effective HPV vaccine programs in Cameroon and other, similar settings.

Objectives The aim of this research project is to evaluate the effectiveness, feasibility, acceptability, and potential for scalability of integrating HPV vaccination into an existing supply- and demand-side sexual and reproductive health and rights (SRHR) intervention to increase HPV vaccine coverage among girls and boys aged 9-13 years in the North and far North regions of Cameroon. The intervention will aim to deliver HPV vaccination through integration with demand- and supply-side program interventions in addition to an existing program implemented by Population Services International-Cameroon (PSI-C) and Association Camerounaise pour le Marketing Social (ACMS): Programme d'Accès aux Services de Santé de la Reproduction (PASSR).

Specific objectives

1. To describe the barriers and facilitators affecting the implementation of HPV vaccination services for VYA girls (aged 9-13) in the North and Far North Regions of Cameroon, and to assess how these impact access and uptake of HPV vaccination.
2. To evaluate the effectiveness of integrating HPV vaccination interventions into existing supply- and demand-side SRHR programs on uptake of HPV vaccination.
3. To evaluate the effectiveness of integrating HPV vaccination interventions into existing supply- and demand-side SRHR programs on uptake of other VYA health service utilization.
4. To assess acceptability, feasibility, cost, equity, and potential for maintenance and scale of HPV vaccination for adolescent girls integrated into an SRHR intervention.
5. To provide evidence for policy integration of HPV vaccine in the adolescent sexual and reproductive health package at the MOH

Methods The study will be conducted in 4 intervention PASSR health districts (HDs) and 4 'standard of care' comparison HDs in the North and Far North regions of Cameroon. It will use a hybrid model of effectiveness and implementation research, with research conducted from approval until December 2025 (with the potential for ongoing data analysis, manuscript preparation, and dissemination through conferences and publications after this end date). Phase 1, the rapid formative and design phase, research activities will include interviews with key informants and secondary analysis of service statistics and program monitoring data. Key informant interview data will contribute to the development of the implementation model, which will also be informed by programmatic co-design workshops. The second phase (implementation) will include a quasi-experimental effectiveness study comparing HPV vaccine administration to girls and boys aged 9-13 years in the intervention and comparison areas, as well as implementation research activities to assess uptake, reach, implementation, activity-based costing and readiness for integration and scale-up. In addition, phase 2 will include analyses of acceptability, feasibility, and satisfaction, using data from key informant interviews; and quantitative exit interviews, focus group discussions, and qualitative in-depth interviews with girls, boys, and caregivers and health professionals. A mixed methodology, integrating quantitative and qualitative research methods, will be used.

During the formative phase (phase 1), primary data collection will consist of around forty key informant interviews (KIIs), 20 per implementation region; in addition, a secondary analysis of existing routine data will be carried out. During the implementation phase (phase 2), approximately 40 key informant interviews with key stakeholders and a further 40 in-depth interviews with health workers, girls and boys aged 9-13 affected by the programme and their caregivers (e.g. parents and/or guardians) will be conducted. Exit interviews will be conducted with approximately 400 VYA/caregiver dyads after receiving HPV vaccination services in intervention areas. In addition, anonymized routine monitoring data, including aggregated service delivery data collected from the programme monitoring systems as well as from the Cameroon Ministry of Health's DHIS2 platform (an open source health information management system) and other existing data sources, will be extracted and analyzed in both comparison and intervention sites to assess the effectiveness of the intervention. Costing data will also be collected. No primary data collection proposed in this study will be conducted in comparison health facilities or their catchment areas; routine data from comparison facilities will be extracted from DHIS2 and other routine program monitoring systems only for the purposes of the effectiveness component. Primary quantitative data (e.g. exit interviews) will be collected electronically using structured questionnaires, administered via the Open Data Kit on study devices. Qualitative interviews will be recorded using digital audio recorders.

Descriptive analysis, using frequencies, percentages, cross-tabulations, graphs and multivariate and time series analysis, will be carried out to analyze and present the quantitative data. Qualitative data will be systematically transcribed and analyzed using thematic analysis, in which the data will be structured and analyzed using a hybrid deductive-inductive approach, in which the qualitative data is parsed into codes based on the semi-structured interview guide (deductive) as well as emergent codes (inductive). The study protocol will be reviewed and approved by the Cameroon National Ethics Committee and the Population Services International Research Ethics Board (REB). The content of the consent will be explained verbally and written informed consent/assent will be obtained from all study participants; written parental/guardian consent will also be obtained for all minor participants.

Expected outcomes The expected outcome of this study is to provide evidence of the effectiveness, acceptability and scalability of integrating HPV vaccination into existing SRHR supply- and demand-side programming in order to increase HPV vaccination coverage among girls and boys aged 9-13 years in the North and Far North regions of Cameroon. Qualitative results will provide insight into the acceptability of this approach among caregivers, adolescents and health providers, while assessments of scalability and readiness for integration will provide crucial information on feasibility and cost-effectiveness.

The main results of the study will include data on HPV vaccination and other VYA services among girls and boys aged 9-13 in the intervention and comparison areas. The results of the study will be disseminated at a national workshop and scientific conferences, and the findings THwill be submitted for publication in peer-reviewed journals.

Currently, only phase 1 of this study protocol has been approved. A later review and approval of phase 2 activities will be obtained prior to the commencement of phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Key informant identified by study and implementation teams (purposive sampling by key informant type)

Exclusion Criteria:

* Does not provide written informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
HPV vaccine delivery | The primary outcome measure is an aggregated, facility-level outcome which will be assessed at the facility-month level using aggregated routine service statistics data over a period of up to 36 months
  Number of HPV vaccinations provided to adolescents aged 9-13 years old per facility per month

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Mbacham, ScD, DS, Principal Investigator — Fobang Institutes for Innovations in Science and Technology

IPD SHARING:
Plan to Share IPD: Yes
The primary aim of this study is to evaluate the impact of the intervention on delivery of HPV vaccinations to adolescents in Cameroon. No IPD will be used to evaluate the primary outcome for the effectiveness component of this study; rather, the effectiveness component will be assessed using aggregated service statistics data, which is inherently de-identified. These data will be made publicly available, as will other primary data collected in the study (quantitative exit survey data, which is an anticipated activity under phase 2 which has not yet been approved). Qualitative data, particularly from key informants, may be more difficult to completely de-identify; therefore, the investigators will make the decision during inspection of qualitative interview transcripts as to whether all qualitative data can be de-identified adequately to make pubicly available.
Supporting Information: Study Protocol, ICF